CLINICAL TRIAL: NCT02634502
Title: Radiofrequency Ablation Combined With S-1 for Pancreatic Cancer With Liver Metastasis: Correlation Analysis of Prognosis and microRNA Expression
Brief Title: Radiofrequency Ablation Combined With S-1 for Pancreatic Cancer With Liver Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, Ph D, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFA-2013
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Pancreatic
Keywords: radiofrequency; chemotherapy; microRNA
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiofrequency Ablation; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients will receive radiofrequency ablation for liver metastatic lesions, as well as two weeks of oral S-1 treatment every three weeks, until progression of disease or adverse effects leading to termination of treatment. Each 3-week period is one cycle of treatment.
  Interventions: Procedure: radiofrequency ablation; Drug: S-1

INTERVENTIONS:
Procedure: radiofrequency ablation
Drug: S-1

SUMMARY:
This study aims to explore the efficacy and safety of radiofrequency ablation combined with S-1 in pancreatic cancer patients with liver metastasis, as well as the correlation of serum microRNA and patients' prognosis. This protocol will be overseen by the Fudan University Institutional Review Board which has Federal Wide Assurance through the U.S. Department of Health & Human Services (Approved: April 25, 2002).

DETAILED DESCRIPTION:
Primary Outcome Measures:

To evaluate the overall survival (OS) in pancreatic cancer patients with liver metastasis treated with radiofrequency ablation combined with S-1.

Secondary Outcome Measures:

1. To explore the correlation of OS and serum microRNA of the patients.
2. To evaluate the progression free survival (PFS) and its correlation with serum microRNA.
3. To observe the objective response rate (ORR) and adverse effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Status ≥ 70
* Histologically/cytologically confirmed pancreatic adenocarcinoma.
* Patients must have underwent radical resection of the pancreatic lesion, or have their locally advanced pancreatic lesion controlled after first-line chemotherapy.
* At least one measurable liver metastasis by RECIST criteria must be present.
* Single liver metastasis smaller than 5cm, or multiple liver metastases less than 6 lesions and smaller than 3cm for each, without metastasis to other sites.
* Patients must have adequate organ functions reflected by the laboratory criteria below:

Granulocytes ≥ 2,000/uL, Hemoglobin ≥ 8.0 gm/dL, Platelets ≥ 100,000/uL, Serum creatinine < 2.0 mg/dL, Bilirubin < 1.5 mg/dL, SGPT < 2.5 x normal, prothrombin time <13.5s

* Prior therapy, e.g., chemotherapy, radiation, is allowed provided that at least 4 weeks washout time is given.
* Patients with jaundice must have a biliary drainage decompression operation before recruitment.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior treatment with S-1.
* Liver metastatic lesion is located at the surface of the liver, with more than 1/3 of the tumor protruding outside.
* Subject has Child-Pugh grade Class C hepatic impairment, massive ascites, active gastrointestinal bleeding, severe coagulation disorder that could not be corrected, or other contraindication for radiofrequency ablation.
* Tumor invasion of Cavity organs.
* Known central nervous system involvement and leptomeningeal disease.
* Concurrent infection requiring intravenous antibiotics.
* Other serious illness or condition including cardiac disease including congestive heart failure (New York Heart Association Classification III or IV), active HIV infection/HIV disease, psychiatric disorders.
* Subject has previous or concurrent cancer that is distinct in primary site or histology from pancreatic adenocarcinoma except cervical carcinoma in situ, non-melanoma carcinoma of the skin or in situ carcinoma of the bladder. Any cancer curatively treated greater than 3 years prior to entry is permitted.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death, assessed up to 100 months.

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China